CLINICAL TRIAL: NCT02814656
Title: A Phase I, Single Centre, Randomised, Single Blind, Placebo-Controlled Study to Investigate the Safety, Tolerability and Pharmacokinetics of Multiple Ascending Doses of Inhaled AZD8871 in Healthy Male Subjects
Brief Title: Safety, Tolerability and Pharmacokinetics of Multiple Ascending Doses of AZD8871 in Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Collaborators: Parexel (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: D6640C00003
Record Dates: First submitted 2016-06-16; First posted 2016-06-28 (Estimated); Results first posted 2019-02-15 (Actual); Last update posted 2019-02-15 (Actual); Status verified 2018-09

CONDITIONS: Chronic Obstructive Pulmonary Disease
Keywords: muscarinic receptor antagonist and β2 adrenoceptor agonist [MABA]; chronic obstructive pulmonary disease; Asthma (in combination with an inhaled corticosteroid [ICS]; alpha-lactose monohydrate; dry powder inhaler; long-acting β2-agonist (LABA); long-acting muscarinic antagonist (LAMA); fixed-dose combination (FDC)
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Asthma | interventions — AZD-8871

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (3):
- Cohort 1, AZD8871 300 μg or placebo (Experimental): In Cohort 1, participants will receive a single dose of AZD8871 300 μg or placebo on Day 1, followed by once daily dosing on Days 5 to 16.
  Interventions: Drug: AZD8871; Drug: Placebo
- Cohort 2, AZD8871 600 μg or placebo (Experimental): In Cohort 2, participants will receive a single dose of AZD8871 600 μg or placebo on Day 1, followed by once daily dosing on Days 5 to 16.
  Interventions: Drug: AZD8871; Drug: Placebo
- Cohort 3, AZD8871 900 μg or placebo (Experimental): In Cohort 3, participants will receive a single dose of AZD8871 900 μg or placebo on Day 1, followed by once daily dosing on Days 5 to 16.
  Interventions: Drug: AZD8871; Drug: Placebo

INTERVENTIONS:
Drug: AZD8871 — Multiple inhaled doses of AZD8871 will be administered via single dose dry powder inhaler (DPI). Each subject will receive a single inhaled dose of AZD8871 on Day 1 and then single once daily inhalations of AZD8871 will be administered for 12 days from Day 5 until Day 16.
Drug: Placebo — Multiple inhaled doses of placebo powder will be administered via single dose DPI. Each subject will receive a single inhaled dose of placebo on Day 1 and then single once daily inhalations of placebo will be administered for 12 days from Day 5 until Day 16.

SUMMARY:
AZD8871 is a new chemical entity possessing long-acting effect in a single molecule which presents a novel treatment approach to chronic obstructive pulmonary disease [COPD] and potentially also asthma (in combination with an inhaled corticosteroid [ICS]). The therapeutic goal for AZD8871 is a treatment with greater efficacy than single mechanism bronchodilators, with an equivalent or superior safety and tolerability profile. The primary purpose of this study is to check the safety and tolerability of AZD8871 at steady state. A multiple ascending dose (MAD) design has been selected for this study following the first time in man (FTIM), single ascending dose (SAD) study. Three dose levels will be tested in an ascending manner. The first dose to be administered will be 300 μg and the 2 subsequent doses will be decided based on safety, tolerability and pharmacokinetic (PK) data generated in the previous dose. The aim of this study is to also enable further investigations in healthy subjects to evaluate and develop AZD8871 as a dual action bronchodilator with an acceptable side-effect profile compared to other inhaled bronchodilators on the market as a treatment for COPD and asthma.

DETAILED DESCRIPTION:
AZD8871 is a new chemical entity possessing long-acting dualpharmacology (muscarinic receptor antagonist and β2 adrenoceptor agonist [MABA]) in a single molecule. This type of agent presents a novel approach to the treatment of chronic obstructive pulmonary disease [COPD] and potentially also asthma (in combination with an inhaled corticosteroid [ICS]). AZD8871 is being developed for inhalation, formulated with alpha-lactose monohydrate and delivered by dry powder inhaler (DPI) that allows delivery of a single dose of the study drug. By combining this bi-functional activity, the therapeutic goal for AZD8871 is a treatment with greater efficacy than single mechanism bronchodilators, equivalent to long-acting β2-agonist (LABA) and long-acting muscarinic antagonist (LAMA) administered as free- or fixed-dose combination (FDC) therapies, with an equivalent or superior safety and tolerability profile. The current study will start with a single dose of 300 μg AZD8871 or placebo administered to 8 healthy subjects following a 3-day washout period, dosing will then continue for a further 12 days. Following the 1st cohort, 2 further cohorts of 8 subjects each will be administered multiple ascending doses (MAD) of AZD8871 in the same manner as Cohort 1. A MAD design has been selected for this study following the first time in man (FTIM), single ascending dose (SAD) study. Each subject will only be dosed in 1 cohort. The study design allows a gradual escalation of dose (Cohorts 2 and 3) with intensive safety monitoring to ensure the safety of the subjects. In Cohort 1, subjects will receive a single dose of AZD8871 300 μg or placebo on Day 1, followed by once daily dosing on Days 5 to 16. The dosing schedule of all cohorts will be single dose of IMP (active or placebo) on Day 1, followed by once daily dosing on Days 5 to 16. Within 5 to 7 days of discharge from the unit, there will be a Follow-up Visit. Dosing of Cohorts 2 and 3 will be preceded by a safety review committee (SRC) meeting, which will decide the exact dose to be given in the subsequent cohort. The dose escalation between cohorts will not exceed a multiple of 3 and the AZD8871 dose level in the study, for any cohort, will not exceed 2100 μg per day. The planned dose for Cohort 2 is either 600 or 900 μg, however the SRC may decide a different dose level. A minimum of 5 subjects on active treatment need to complete dosing per cohort in order to proceed to the next dose level. The aim of this study is to also enable further investigations in healthy subjects to evaluate and develop AZD8871 as a dual action bronchodilator with an acceptable side-effect profile compared to other inhaled bronchodilators on the market as a treatment for COPD and asthma.

ELIGIBILITY:
Inclusion Criteria:

1. Provision of written informed consent prior to conducting any study-related procedures, including withdrawal of medications.
2. Male subjects aged 18 to 55 years, inclusive at Screening.
3. Body mass index (BMI) calculated as weight in kg/height in m2 from ≥18 to ≤30 kg/m2 and weight ≥50 kg at Screening.
4. Healthy, free from any clinically significant disease/ conditions (including all cardiovascular conditions), as determined by medical history, physical examination, clinical laboratory testing, 12-lead ECG findings at Screening and admission to the unit.
5. Spirometry readings (FEV1 and Forced Vital Capacity [FVC]) to be ≥80% of predicted value calculated using Quanjer 2012 reference equations (Quanjer et al 2012) at Screening.
6. Normal blood pressure (BP) (defined as systolic BP [SBP] ≥90 and ≤140 mmHg, and diastolic BP [DBP] ≥50 and ≤90 mmHg) at Screening and admission to the unit, measured after resting in supine position for at least 10 minutes.
7. Normal heart rate (HR) (defined as HR ≥45 and ≤90) measured after resting in supine position for at least 10 minutes at Screening and admission to the unit.
8. Negative for hepatitis B surface antigen (HBsAg), hepatitis B core (HBc) antibody (IgM), hepatitis C antibody and human immunodeficiency virus (HIV) I and II antibodies at Screening.
9. Negative for drugs of abuse and alcohol tests at Screening and admission to the unit.
10. Normal serum potassium at Screening and at admission to the unit.
11. Willing and able to comply with study specific procedures and restrictions

Exclusion Criteria:

1. Involvement in the planning and/or conduct of the study (applies to both AstraZeneca staff and/or staff at the study site).
2. Surgical history clinically relevant for the purpose of the study or any clinically significant illness, medical/surgical procedure or trauma within 4 weeks of Screening.
3. History of malignancy of any organ system, treated or untreated within the past 5 years, with the exception of localised basal cell carcinoma of the skin.
4. Current smokers, or a smoking history during the last 6 months or total smoking history of more than 10 pack-years. Use of electronic cigarettes or other forms of nicotine, current use or use within the last 6 months.
5. Prolonged QTcF interval, >450 ms at Screening, or family history of long QT syndrome.
6. Any clinically significant arrhythmia noted on telemetry recording, prior to randomisation.
7. History of excessive use or abuse of alcohol within the past 2 years.
8. History of drug abuse within the past 2 years.
9. Donation or loss >400 ml of blood and plasma within the previous 3 months prior to Visit 1, Screening.
10. History of presence of severe allergy/hypersensitivity or ongoing allergy/hypersensitivity to any drug, as judged by the Investigator or history of hypersensitivity to drugs pharmacologically related to study drug.
11. PR (PQ) interval shortening <120 ms (PR >110 ms but <120 ms is acceptable if there is no evidence of ventricular pre-excitation) at Screening.
12. PR (PQ) interval prolongation (> 240 ms), intermittent second (Wenckebach block while asleep is not exclusive), or third degree atrioventricular block, or atrioventricular dissociation at Screening.
13. Persistent or intermittent complete bundle branch block (BBB), incomplete bundle branch block (IBBB), or intraventricular conduction delay (IVCD) with QRS >110 ms.
14. Subject who does not agree to follow instructions to avoid partner pregnancy.
15. Subject who is not able to adhere to the restrictions on prior and concomitant medications.
16. Used any investigational drug within 3 months prior to Screening or within the equivalent time of 5 half-lives of receiving the last administration, whichever is longer, or on an extended follow-up after receiving an IMP.
17. Subjects unable to communicate reliably with the Investigator.
18. Vulnerable subjects, e.g., kept in detention, protected adults under guardianship, trusteeship, or committed to an institution by governmental or juridical order.

Ages: 18 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2016-06-22 (Actual); Primary Completion 2016-11-28 (Actual); Study Completion 2016-11-28 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Muna Albayaty, MBChB, MSc, MFPM, Principal Investigator — Parexel
Locations (1):
- Research Site, London, United Kingdom

REFERENCES:
- [Derived] Balaguer V, Albayaty M, Jimenez E, Wahlby-Hamren U, Astbury C, Seoane B, Malice MP, Lei A, Aggarwal A, Psallidas I. Navafenterol (AZD8871) in healthy volunteers: safety, tolerability and pharmacokinetics of multiple ascending doses of this novel inhaled, long-acting, dual-pharmacology bronchodilator, in two phase I, randomised, single-blind, placebo-controlled studies. Respir Res. 2020 Sep 9;21(Suppl 1):212. doi: 10.1186/s12931-020-01474-1. PMID 32907575

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study was conducted at a single centre in the UK. The first patient was screened in June 2016 and the last patient visit was in November 2016.
Pre-assignment Details: A single dose of 300 μg AZD8871 or placebo was administered to 8 healthy subjects following a 3-day washout period, dosing then continued for a further 12 days. Following the 1st cohort, 2 further cohorts of 8 subjects each were administered multiple ascending doses of AZD8871 in the same manner as Cohort 1.
Groups:
- 300 μg AZD8871: Participants received a single dose of AZD8871 300 μg on Day 1, followed by once daily dosing on Days 5 to 16.
- 600 μg AZD8871: Participants received a single dose of 600 μg AZD8871 on Day 1, followed by once daily dosing on Days 5 to 16.
- 900 μg AZD8871: Participants received a single dose of 900 μg AZD8871 on Day 1, followed by once daily dosing on Days 5 to 16.
- Placebo: Participants received a single dose of Placebo on Day 1, followed by once daily dosing on Days 5 to 16.
Period: Overall Study
Arm/Group | 300 μg AZD8871 | 600 μg AZD8871 | 900 μg AZD8871 | Placebo
Started | 6 | 6 | 6 | 6
Completed | 6 | 6 | 6 | 6
Not Completed | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | 300 μg AZD8871 | 600 μg AZD8871 | 900 μg AZD8871 | Placebo | Total
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 24
Age, Continuous [Mean (Standard Deviation); unit: Years] | 34.0 (5.7) | 44.2 (7.9) | 36.5 (6.8) | 41.5 (7.6) | 39.0 (7.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0 | 0 | 0
  Male | 6 | 6 | 6 | 6 | 24

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With ≥1 Treatment Emergent Adverse Event in Any Category.
Description: Recording treatment emergent adverse events (TEAE).
  A TEAE was defined as an AE with onset (start date/time) after the first dose of investigational medicinal product. An AE is the development of an undesirable medical condition or the deterioration of a pre-existing medical condition following or during exposure to a pharmaceutical product, whether or not considered causally related to the product. An undesirable medical condition can be symptoms (e.g., nausea, chest pain), signs (e.g., tachycardia, enlarged liver) or the abnormal results of an investigation (e.g., laboratory findings, ECG).
Time Frame: Change from baseline up to Days 25-27
Population: Safety analysis population: defined as all participants who received at least one dose of the investigational product and for whom any post-dose safety data were available.
Measure: Count of Participants; unit: Participants
Arm/Group | 300 μg AZD8871 | 600 μg AZD8871 | 900 μg AZD8871 | Placebo
Number analyzed (Participants) | 6 | 6 | 6 | 6
Participants | 3 | 1 | 5 | 4

2. Secondary Outcome: Observed Maximum Concentration (Cmax) of AZD8871 and Its Metabolites (Single Dose).
Description: Observed maximum concentration, taken directly from the individual concentration-time curve (Cmax) of AZD8871 and its metabolites (LAS191861 and LAS34850).
Time Frame: Day 1, pre-dose and at 15, 30 and 45 minutes and 1, 1.5, 2, 3, 4, 6, 8, 12, 16, 24, 36, 48, 72 and 96 hours post-dose
Population: Pharmacokinetic analysis population: defined as all participants in the safety analysis population who received at least 1 dose of AZD8871 and had at least 1 of the parameters Cmax, AUC or AUClast evaluable for AZD8871 and were assumed not to be affected by factors such as protocol deviations.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: pg/mL
Arm/Group | 300 μg AZD8871 | 600 μg AZD8871 | 900 μg AZD8871 | Placebo
Number analyzed (Participants) | 6 | 6 | 6 | 0
pg/mL
  AZD8871: number analyzed (Participants) | 6 | 5 | 6 | 0
  AZD8871 | 397.0 (28.66) | 991.1 (63.45) | 1568 (20.41) |
  LAS191861: number analyzed (Participants) | 6 | 5 | 6 | 0
  LAS191861 | 20.17 (28.38) | 60.08 (50.10) | 96.31 (24.66) |
  LAS34850: number analyzed (Participants) | 6 | 5 | 6 | 0
  LAS34850 | 708.5 (31.44) | 1376 (19.63) | 1839 (33.17) |

3. Secondary Outcome: Observed Maximum Concentration (Cmax) of AZD8871 and Its Metabolites (Day 16).
Description: as for outcome 2
Time Frame: Day 16, pre-dose and at 15, 30 and 45 minutes and 1, 1.5, 2, 3, 4, 6, 8, 12, 16, 24, 36, 48, 72 and 96 hours post-dose
Population: as for outcome 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: pg/mL
Arm/Group | 300 μg AZD8871 | 600 μg AZD8871 | 900 μg AZD8871 | Placebo
Number analyzed (Participants) | 6 | 6 | 6 | 0
pg/mL
  AZD8871 | 406.5 (34.44) | 1018 (53.64) | 1830 (28.47) |
  LAS191861 | 53.80 (35.18) | 119.3 (39.47) | 204.5 (25.14) |
  LAS34850 | 905.4 (29.90) | 2067 (21.49) | 2340 (38.41) |

4. Secondary Outcome: Time to Reach Maximum Concentration (Tmax) of AZD8871 and Its Metabolites (Single Dose).
Description: Time to reach maximum concentration, taken directly from the individual concentration-time curve (tmax) of AZD8871 and its metabolites (LAS191861 and LAS34850).
Time Frame: Day 1, pre-dose and at 15, 30 and 45 minutes and 1, 1.5, 2, 3, 4, 6, 8, 12, 16, 24, 36, 48, 72 and 96 hours post-dose
Population: as for outcome 2
Measure: Median (Full Range); unit: h
Arm/Group | 300 μg AZD8871 | 600 μg AZD8871 | 900 μg AZD8871 | Placebo
Number analyzed (Participants) | 6 | 6 | 6 | 0
h
  AZD8871: number analyzed (Participants) | 6 | 5 | 6 | 0
  AZD8871 | 1.50 [1.00 to 1.52] | 1.52 [1.50 to 1.55] | 1.51 [1.48 to 1.52] |
  LAS191861: number analyzed (Participants) | 6 | 5 | 6 | 0
  LAS191861 | 1.51 [1.50 to 2.00] | 1.55 [1.50 to 2.02] | 2.00 [1.48 to 2.02] |
  LAS34850: number analyzed (Participants) | 6 | 5 | 6 | 0
  LAS34850 | 4.00 [3.00 to 6.00] | 3.00 [3.00 to 4.02] | 4.00 [2.00 to 5.98] |

5. Secondary Outcome: Time to Reach Maximum Concentration (Tmax) of AZD8871 and Its Metabolites (Day 16).
Description: as for outcome 4
Time Frame: Day 16, pre-dose and at 15, 30 and 45 minutes and 1, 1.5, 2, 3, 4, 6, 8, 12, 16, 24, 36, 48, 72 and 96 hours post-dose
Population: as for outcome 2
Measure: Median (Full Range); unit: h
Arm/Group | 300 μg AZD8871 | 600 μg AZD8871 | 900 μg AZD8871 | Placebo
Number analyzed (Participants) | 6 | 6 | 6 | 0
h
  AZD8871 | 1.50 [1.50 to 1.53] | 1.50 [1.48 to 1.50] | 1.50 [1.50 to 1.50] |
  LAS191861 | 1.50 [1.00 to 2.00] | 1.50 [1.48 to 2.00] | 1.50 [1.50 to 1.50] |
  LAS34850 | 3.51 [1.50 to 4.03] | 4.01 [2.98 to 6.00] | 4.01 [2.00 to 6.00] |

6. Secondary Outcome: Terminal Half-life (t½λz) of AZD8871 and Its Metabolites (Single Dose).
Description: Terminal elimination half-life (t½λz) of AZD8871 and its metabolites (LAS191861 and LAS34850), estimated as (ln2)/ λz.
Time Frame: Day 1, pre-dose and at 15, 30 and 45 minutes and 1, 1.5, 2, 3, 4, 6, 8, 12, 16, 24, 36, 48, 72 and 96 hours post-dose
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: h
Arm/Group | 300 μg AZD8871 | 600 μg AZD8871 | 900 μg AZD8871 | Placebo
Number analyzed (Participants) | 6 | 6 | 6 | 0
h
  AZD8871: number analyzed (Participants) | 6 | 5 | 6 | 0
  AZD8871 | 50.44 (6.796) | 42.89 (11.99) | 49.24 (9.055) |
  LAS191861: number analyzed (Participants) | 4 | 3 | 3 | 0
  LAS191861 | 46.51 (22.36) | 67.90 (57.19) | 69.43 (7.989) |
  LAS34850: number analyzed (Participants) | 6 | 5 | 4 | 0
  LAS34850 | 12.15 (6.649) | 36.37 (21.94) | 37.01 (16.91) |

7. Secondary Outcome: Terminal Half-life (t½λz) of AZD8871 and Its Metabolites (Day 16).
Description: Terminal elimination half-life (t½λz) of AZD8871 and its metabolites (LAS191861 and LAS34850), estimated as (ln2)/ λz.
Time Frame: Day 16, pre-dose and at 15, 30 and 45 minutes and 1, 1.5, 2, 3, 4, 6, 8, 12, 16, 24, 36, 48, 72 and 96 hours post-dose
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: h
Arm/Group | 300 μg AZD8871 | 600 μg AZD8871 | 900 μg AZD8871 | Placebo
Number analyzed (Participants) | 6 | 6 | 6 | 0
h
  AZD8871: number analyzed (Participants) | 6 | 5 | 5 | 0
  AZD8871 | 78.51 (11.01) | 62.39 (16.69) | 70.19 (4.144) |
  LAS191861: number analyzed (Participants) | 1 | 3 | 0 | 0
  LAS191861 | 0.00 (0.00) | 98.78 (30.75) |  |
  LAS34850: number analyzed (Participants) | 5 | 6 | 3 | 0
  LAS34850 | 51.20 (9.373) | 67.07 (27.46) | 61.46 (8.128) |

8. Secondary Outcome: AUC(0-24) of AZD8871 and Its Metabolites (Single Dose).
Description: Area under the plasma concentration-curve from time zero to 24 hours post-dose (AUC[0-24]) of AZD8871 and its metabolites (LAS191861 and LAS34850).
Time Frame: Day 1, pre-dose and at 15, 30 and 45 minutes and 1, 1.5, 2, 3, 4, 6, 8, 12, 16, 24, 36, 48, 72 and 96 hours post-dose
Population: as for outcome 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: pg.h/mL
Arm/Group | 300 μg AZD8871 | 600 μg AZD8871 | 900 μg AZD8871 | Placebo
Number analyzed (Participants) | 6 | 6 | 6 | 0
pg.h/mL
  AZD8871: number analyzed (Participants) | 6 | 5 | 6 | 0
  AZD8871 | 1272 (18.69) | 3805 (58.72) | 4862 (15.58) |
  LAS191861: number analyzed (Participants) | 6 | 5 | 6 | 0
  LAS191861 | 152.5 (20.04) | 493.7 (42.75) | 770.3 (33.90) |
  LAS34850: number analyzed (Participants) | 6 | 5 | 6 | 0
  LAS34850 | 5761 (34.07) | 12540 (23.58) | 18720 (32.55) |

9. Secondary Outcome: AUC(0-24) of AZD8871 and Its Metabolites (Day 16).
Description: as for outcome 8
Time Frame: Day 16, pre-dose and at 15, 30 and 45 minutes and 1, 1.5, 2, 3, 4, 6, 8, 12, 16, 24, 36, 48, 72 and 96 hours post-dose
Population: as for outcome 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: pg.h/mL
Arm/Group | 300 μg AZD8871 | 600 μg AZD8871 | 900 μg AZD8871 | Placebo
Number analyzed (Participants) | 6 | 6 | 6 | 0
pg.h/mL
  AZD8871: number analyzed (Participants) | 6 | 5 | 6 | 0
  AZD8871 | 2103 (25.20) | 5508 (47.25) | 7077 (19.87) |
  LAS191861 | 528.9 (15.70) | 1248 (34.57) | 1911 (34.68) |
  LAS34850 | 8848 (23.82) | 22580 (29.69) | 27300 (28.27) |

10. Secondary Outcome: AUC of AZD8871 and Its Metabolites (Single Dose).
Description: Area under the concentration-time curve of AZD8871 and its metabolites (LAS191861 and LAS34850) from time zero extrapolated to infinity.
  AUC is estimated by AUC0-last + Clast/λz where Clast is the last observed quantifiable concentration.
Time Frame: Day 1, pre-dose and at 15, 30 and 45 minutes and 1, 1.5, 2, 3, 4, 6, 8, 12, 16, 24, 36, 48, 72 and 96 hours post-dose
Population: as for outcome 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: pg.h/mL
Arm/Group | 300 μg AZD8871 | 600 μg AZD8871 | 900 μg AZD8871 | Placebo
Number analyzed (Participants) | 6 | 6 | 6 | 0
pg.h/mL
  AZD8871: number analyzed (Participants) | 6 | 4 | 6 | 0
  AZD8871 | 2218 (21.18) | 5574 (79.73) | 7496 (14.24) |
  LAS191861: number analyzed (Participants) | 0 | 1 | 0 | 0
  LAS191861 |  | 0.00 (0.00) |  |
  LAS34850: number analyzed (Participants) | 6 | 5 | 4 | 0
  LAS34850 | 6553 (38.03) | 16830 (36.65) | 24340 (38.79) |

11. Secondary Outcome: Apparent Clearance for Parent Drug (CL/F) (Single Dose).
Description: Apparent clearance for parent drug (CL/F) estimated as dose divided by AUC of AZD8871.
Time Frame: Day 1, pre-dose and at 15, 30 and 45 minutes and 1, 1.5, 2, 3, 4, 6, 8, 12, 16, 24, 36, 48, 72 and 96 hours post-dose
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: L/h
Arm/Group | 300 μg AZD8871 | 600 μg AZD8871 | 900 μg AZD8871 | Placebo
Number analyzed (Participants) | 6 | 6 | 6 | 0
L/h | 137.8 (28.30) | 133.7 (115.1) | 121.1 (17.47) |

12. Secondary Outcome: Apparent Clearance for Parent Drug (CL/F) (Day 16).
Description: Apparent clearance for parent drug (CL/F) estimated as dose divided by AUC(0-24) of AZD8871.
Time Frame: Day 16, pre-dose and at 15, 30 and 45 minutes and 1, 1.5, 2, 3, 4, 6, 8, 12, 16, 24, 36, 48, 72 and 96 hours post-dose
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: L/h
Arm/Group | 300 μg AZD8871 | 600 μg AZD8871 | 900 μg AZD8871 | Placebo
Number analyzed (Participants) | 6 | 6 | 6 | 0
L/h | 146.2 (33.62) | 120.2 (67.93) | 129.3 (26.27) |

13. Secondary Outcome: Apparent Volume of Distribution for Parent Drug at Terminal Phase (Vz/F) (Single Dose).
Description: Apparent volume of distribution for parent drug at terminal phase (Vz/F) (extravascular administration), estimated by dividing the apparent clearance (CL/F) by λz of AZD8871.
Time Frame: Day 1, pre-dose and at 15, 30 and 45 minutes and 1, 1.5, 2, 3, 4, 6, 8, 12, 16, 24, 36, 48, 72 and 96 hours post-dose
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: L
Arm/Group | 300 μg AZD8871 | 600 μg AZD8871 | 900 μg AZD8871 | Placebo
Number analyzed (Participants) | 6 | 6 | 6 | 0
L | 9873 (1677) | 6737 (4406) | 8724 (2770) |

14. Primary Outcome: Number of Participants With Clinically Relevant Abnormalities in Recording of Physical Examination.
Description: A full physical examination included the examination of the following: general appearance, eyes, ears, nose, throat, chest/respiratory, heart/cardiovascular, gastrointestinal/liver, musculoskeletal/extremities, dermatological/skin, thyroid/neck, lymph nodes, neurological/psychiatric.
  A brief physical examination included assessment of the following: skin, lungs, cardiovascular system and abdomen (liver and spleen).
  A complete physical examination was performed at the Screening Visit. Any abnormal finding assessed as the investigator as clinically relevant was reported as an adverse event.
Time Frame: Change from baseline up to Days 25-27
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | 300 μg AZD8871 | 600 μg AZD8871 | 900 μg AZD8871 | Placebo
Number analyzed (Participants) | 6 | 6 | 6 | 6
Participants | 1 | 0 | 1 | 1

15. Primary Outcome: Number of Participants With Clinically Relevant Abnormalities in Vital Signs (Pulse, Blood Pressure and Body Temperature).
Description: Systolic and diastolic BP (SBP/DBP) (in mmHg) measured after at least 10 minutes (could be reduced to 5 minutes at collection time points within the 1st hour after dosing) resting, and also before taking any blood sample and conducting any spirometry. Measurements were carried out with subject in the supine position and preferably always on the same arm.
  Subject's oral body temperature was measured at each vital signs collection.
Time Frame: Change from baseline up to Days 25-27
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | 300 μg AZD8871 | 600 μg AZD8871 | 900 μg AZD8871 | Placebo
Number analyzed (Participants) | 6 | 6 | 6 | 6
Participants | 0 | 1 | 1 | 1

16. Primary Outcome: Number of Participants With Clinically Relevant New Findings or Worsening of Pre-existing Findings as Assessed by Haematology.
Description: Haematocrit, haemoglobin, erythrocytes (red blood cells), mean corpuscular volume, mean corpuscular haemoglobin, mean corpuscular haemoglobin concentration, leucocytes (white blood cells), differential blood count (neutrophils, lymphocytes, monocytes, eosinophils and basophils), and thrombocytes (platelets).
Time Frame: Changes from baseline up to Days 25-27
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | 300 μg AZD8871 | 600 μg AZD8871 | 900 μg AZD8871 | Placebo
Number analyzed (Participants) | 6 | 6 | 6 | 6
Participants | 0 | 0 | 0 | 0

17. Primary Outcome: Number of Participants With Clinically Relevant Abnormalities in 12-lead Safety ECG.
Description: A 12-lead ECG was obtained after the subject rested in the supine position for at least 10 minutes (could be reduced to 5 minutes at collection time points within the first hour after dosing) (using the sites own ECG machines when not performing dECGs and using the same machine as the dECGs when time points coincided).
Time Frame: Changes from baseline up to Days 25-27
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | 300 μg AZD8871 | 600 μg AZD8871 | 900 μg AZD8871 | Placebo
Number analyzed (Participants) | 6 | 6 | 6 | 6
Participants | 0 | 0 | 0 | 0

18. Primary Outcome: Number of Participants With Clinically Relevant Abnormalities in Telemetry ECG.
Description: Recording of telemetry findings. A 2-lead real-time telemetry ECG was performed for at least 4 hours on Day -1 and then on Days 1, 10 and 16 from 30 minutes pre-dose until 24 hours post-dose. The telemetry monitoring system was reviewed by the Investigator or research nurse and paper printouts of any clinically important events were stored as source data.
Time Frame: Changes from baseline up to Day 20 (discharge from study unit)
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | 300 μg AZD8871 | 600 μg AZD8871 | 900 μg AZD8871 | Placebo
Number analyzed (Participants) | 6 | 6 | 6 | 6
Participants | 0 | 0 | 0 | 0

19. Primary Outcome: Number of Participants With Clinically Relevant New Findings or Worsening of a Pre-existing Findings as Assessed by Clinical Chemistry.
Description: Electrolytes: Sodium, potassium, calcium, chloride and inorganic phosphorus Enzymes: AST, ALT, ALP, GGT, LDH, creatine-kinase Substrates: Glucose (fasting), total cholesterol, triglycerides, creatinine, TBL, total protein, albumin, uric acid, urea and BUN Endocrinology: T4, TSH Viral Serology: HIV I and II antibodies, Hepatitis C antibodies, Hepatitis B surface antigen, Hepatitis B core (HBc) immunoglobulin antibodies Coagulation parameters: INR, PT, aPTT
Time Frame: Changes from baseline up to Days 25-27
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | 300 μg AZD8871 | 600 μg AZD8871 | 900 μg AZD8871 | Placebo
Number analyzed (Participants) | 6 | 6 | 6 | 6
Participants | 0 | 0 | 0 | 0

20. Primary Outcome: Number of Participants With Clinically Relevant New Findings or Worsening of Pre-existing Findings as Assessed by Urinalysis Report.
Description: Dipstick analysis was performed at the centre and included: pH, blood, leucocytes, protein, glucose, bilirubin, urobilinogen, ketones and nitrites. If clinically relevant abnormalities were detected (positive result in dipstick), microscopy (RBC, WBC and casts [Hyaline, Granular and Cellular]) were performed.
Time Frame: Changes from baseline up to Days 25-27
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | 300 μg AZD8871 | 600 μg AZD8871 | 900 μg AZD8871 | Placebo
Number analyzed (Participants) | 6 | 6 | 6 | 6
Participants | 0 | 0 | 0 | 0

21. Primary Outcome: Number of Participants With Clinically Relevant Abnormalities in 12-lead dECG (Including High Precision QTc Analysis) Findings.
Description: The AZ ECG Centre performed the digital ECG (dECG) analysis in this study, using the EClysis© system, version 3.3, or higher. At protocol-indicated time points, 12-lead continuous dECG was recorded over at least 5 minutes with the Schiller Cardiovit CS-200 recorder (Schiller AG, Baar, Switzerland) and transmitted to the AZ central dECG repository, according to AZ ECG Centre´s standard procedures for settings, recording and transmission of dECGs
Time Frame: Changes from baseline up to Day 20
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | 300 μg AZD8871 | 600 μg AZD8871 | 900 μg AZD8871 | Placebo
Number analyzed (Participants) | 6 | 6 | 6 | 6
Participants | 0 | 0 | 0 | 0

22. Secondary Outcome: Accumulation Ratio for Cmax (Rac[Cmax]) for AZD8871 and Its Metabolites (Day 16).
Description: Accumulation ratio for Cmax estimated as (Cmax pg/mL on Day 16/ Cmax pg/mL on Day 1) of AZD8871 and its metabolites (LAS191861 and LAS34850).
Time Frame: Days 1 and 16, pre-dose and at 15, 30 and 45 minutes and 1, 1.5, 2, 3, 4, 6, 8, 12, 16, 24, 36, 48, 72 and 96 hours post-dose
Population: as for outcome 2
Measure: Mean (Full Range); unit: Ratio
Arm/Group | 300 μg AZD8871 | 600 μg AZD8871 | 900 μg AZD8871 | Placebo
Number analyzed (Participants) | 6 | 6 | 6 | 0
Ratio
  AZD8871: number analyzed (Participants) | 6 | 5 | 6 | 0
  AZD8871 | 1.032 [0.881 to 1.23] | 1.054 [0.979 to 1.12] | 1.181 [0.843 to 1.40] |
  LAS191861: number analyzed (Participants) | 6 | 5 | 6 | 0
  LAS191861 | 2.794 [1.79 to 4.77] | 1.897 [1.59 to 2.04] | 2.153 [1.67 to 2.70] |
  LAS34850: number analyzed (Participants) | 6 | 5 | 6 | 0
  LAS34850 | 1.304 [1.00 to 1.67] | 1.431 [1.30 to 1.51] | 1.275 [1.19 to 1.44] |

23. Secondary Outcome: Accumulation Ratio for AUC0-24 (Rac[AUC0-24]) for AZD8871 and Its Metabolites (Day 16).
Description: Accumulation ratio for AUC0-24 (Rac[AUC0-24]) for AZD8871 and its metabolites (LAS191861 and LAS34850) estimated as (AUC(0-24) pg.h/mL on Day 16/ AUC(0-24) pg.h/mL on Day 1).
Time Frame: as for outcome 22
Population: as for outcome 2
Measure: Mean (Full Range); unit: Ratio
Arm/Group | 300 μg AZD8871 | 600 μg AZD8871 | 900 μg AZD8871 | Placebo
Number analyzed (Participants) | 6 | 6 | 6 | 0
Ratio
  AZD8871: number analyzed (Participants) | 6 | 5 | 6 | 0
  AZD8871 | 1.675 [1.33 to 2.14] | 1.451 [1.25 to 1.60] | 1.463 [1.20 to 1.58] |
  LAS191861: number analyzed (Participants) | 6 | 5 | 6 | 0
  LAS191861 | 3.510 [2.55 to 4.28] | 2.398 [1.83 to 3.08] | 2.494 [2.20 to 3.00] |
  LAS34850: number analyzed (Participants) | 6 | 5 | 6 | 0
  LAS34850 | 1.564 [1.22 to 2.04] | 1.690 [1.55 to 1.90] | 1.463 [1.23 to 1.55] |

ADVERSE EVENTS:
Time Frame: From baseline to the Follow-up Visit at Days 25-27
Description: The safety analysis population included all subjects who received at least 1 dose of the investigational product and for whom any post-dose safety data were available.
Arm/Group | 300 μg AZD8871 | 600 μg AZD8871 | 900 μg AZD8871 | Placebo
All-Cause Mortality (participants affected / at risk) | 0/6 | 0/6 | 0/6 | 0/6
Serious Adverse Events (participants affected / at risk) | 0/6 | 0/6 | 0/6 | 0/6
Other Adverse Events (participants affected / at risk) | 3/6 | 1/6 | 5/6 | 4/6
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 300 μg AZD8871 (N=6) | 600 μg AZD8871 (N=6) | 900 μg AZD8871 (N=6) | Placebo (N=6)
Vessel puncture site bruise (General disorders) | 0 (0) | 0 (0) | 3 (3) | 2 (2)
Vessel puncture site pain (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Headache (Nervous system disorders) | 2 (2) | 1 (1) | 0 (0) | 0 (0)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Toothache (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Nasopharyngitis (Infections and infestations) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Contact dermatitis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Dry skin (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Arthropod sting (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Publication and / or presentation whether complete or partial, of any part of the data or results of this study will not be allowed until global publication and study results disclosure by the sponsor as per EMA / FDA regulatory compliance obligations, and only after mutual agreement between the Investigator and AstraZeneca